CLINICAL TRIAL: NCT06086587
Title: Development and Application of Molecular Evaluation Instrument for Lung Cancer Diagnosis and Treatment
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Yayi He, Principal Investigator, Shanghai Pulmonary Hospital, Shanghai, China
Other Study IDs: 2022tjdxsy048
Record Dates: First submitted 2023-09-26; First posted 2023-10-17 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The precise diagnosis and treatment of lung cancer is not only a major national strategic need but also an urgent demand from the general public. The "three stages" of precise diagnosis and treatment of lung cancer include early diagnosis, effective treatment, and precise evaluation. Currently, invasive methods are mainly used in these three stages of clinical practice. The non-invasive molecular diagnosis of early-stage lung cancer and the molecular evaluation of treatment efficacy are critical core issues in lung cancer clinical diagnosis and treatment. In response to this problem, this project aims to use exhaled breath as a sample to develop a scientific instrument with independent intellectual property rights, which integrates early-stage diagnosis of lung cancer and evaluation of treatment efficacy. We will also conduct related application research to meet the needs of the public and contribute to the health of the entire population.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participate in the clinical study; fully understand and be informed about this study, and sign the informed consent form (ICF); willing to comply with and have the ability to complete all trial procedures.
2. Male or female participants aged 18-75 (inclusive) at the time of signing the ICF.
3. The case group included patients diagnosed with lung cancer, including early-stage and advanced-stage patients; the control group consisted of healthy individuals without a history of lung cancer or related respiratory diseases.
4. At least one measurable target lesion evaluated according to RECIST 1.1 criteria by the Institutional Review and Research Committee (IRRC).
5. Patients provide eligible tumor tissue for histopathological testing as required.
6. Relevant laboratory tests indicate tolerance to chemotherapy and immunotherapy.

Exclusion Criteria:

1. Patients with unclear diagnosis of lung cancer.
2. Patients with contraindications to chemotherapy or immunotherapy.
3. Patients with contraindications to lung tissue examination.
4. Patients with other respiratory diseases within the year or concurrent respiratory system diseases (such as chronic obstructive pulmonary disease, bronchial asthma, etc.).
5. Patients with other active malignant tumors within the year or concurrently.
6. Patients with severe heart disease and patients with other severe diseases (such as liver dysfunction, renal dysfunction, etc.).
7. Patients known to have a history of psychiatric drug abuse or drug addiction; patients with a history of alcohol abuse.
8. Based on the investigator's judgment, patients have other factors that may lead to premature termination of this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Biopsy patients in Shanghai Pulmonary Hospital
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-11-07 (Estimated); Primary Completion 2024-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
OS | From date of diagnosis until the date of death from any cause, whichever came first, assessed up to 24 months
  Time from randomization to death (from any cause)
PFS | From date of diagnosis until the date of first documented progression from any cause, whichever came first, assessed up to 24 months
  The time between the initiation of randomization and the occurrence (any aspect) of tumor progression or death (from any cause)
ORR | The proportion of patients who achieved a 30%(usual) reduction in tumor volume while maintaining the minimum required duration was calculated at month 24 of the study
  Refers to the proportion of subjects whose tumors shrink by a certain amount and remain for a certain period of time, including those with CR+PR
DOR | The time from first diagnosis of CR or PR to diagnosis of PD was calculated at 24 months of study
  Is the time from the first documented response (CR or PR) to the first documented disease progression or death, whichever occurs first

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carozzi FM, Bisanzi S, Carrozzi L, Falaschi F, Lopes Pegna A, Mascalchi M, Picozzi G, Peluso M, Sani C, Greco L, Ocello C, Paci E; ITALUNG Working Group. Multimodal lung cancer screening using the ITALUNG biomarker panel and low dose computed tomography. Results of the ITALUNG biomarker study. Int J Cancer. 2017 Jul 1;141(1):94-101. doi: 10.1002/ijc.30727. Epub 2017 Apr 21. PMID 28387927
- [Background] Kusano M, Mendez E, Furton KG. Development of headspace SPME method for analysis of volatile organic compounds present in human biological specimens. Anal Bioanal Chem. 2011 Jun;400(7):1817-26. doi: 10.1007/s00216-011-4950-2. Epub 2011 Apr 6. PMID 21598081
- [Background] Jones AW, Lagesson V, Tagesson C. Determination of isoprene in human breath by thermal desorption gas chromatography with ultraviolet detection. J Chromatogr B Biomed Appl. 1995 Oct 6;672(1):1-6. doi: 10.1016/0378-4347(95)00207-y. PMID 8590920
- [Background] Bruderer T, Gaisl T, Gaugg MT, Nowak N, Streckenbach B, Muller S, Moeller A, Kohler M, Zenobi R. On-Line Analysis of Exhaled Breath Focus Review. Chem Rev. 2019 Oct 9;119(19):10803-10828. doi: 10.1021/acs.chemrev.9b00005. Epub 2019 Aug 21. PMID 31594311
- [Background] Zou Y, Zhang X, Chen X, Hu Y, Ying K, Wang P. Optimization of volatile markers of lung cancer to exclude interferences of non-malignant disease. Cancer Biomark. 2014;14(5):371-9. doi: 10.3233/CBM-140418. PMID 25171479